CLINICAL TRIAL: NCT06107608
Title: Molecular Imaging of FAP Expressing Cancer-associated Fibroblasts in NSCLC Treated With Immune-checkpoint Inhibitors
Acronym: LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-MN-LIFE1
Record Dates: First submitted 2023-09-26; First posted 2023-10-30 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Immunotherapy; FAPI-46; Non Small Cell Lung Cancer; PET; PET/CT; fibroblast activation protein; fibroblast activation protein inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: molecular imaging of FAP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAPI PET/CT (Experimental): The radiopharmaceutical 68Gallium-FAPI-46 (FAPI) is injected intravenously for molecular imaging of FAP expression with FAPI PET/CT in patients with NSCLC with an indication for immunotherapy
  Interventions: Procedure: FAPI PET/CT

INTERVENTIONS:
Procedure: FAPI PET/CT — The radiopharmaceutical 68Gallium-FAPI-46 (FAPI) is injected intravenously for molecular imaging of FAP expression with FAPI PET/CT.

SUMMARY:
Evaluation of the relation between baseline fibroblast activation protein (FAP) expression based on Ga-FAPI uptake with patient outcome among NSCLC patients receiving immunotherapy for recurrent/metastatic disease.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP), a type II membrane glycoprotein, is selectively expressed by cancer-associated fibroblasts (CAFs) in more than 90% of epithelial carcinomas. FAP also regulates antitumor immune response. For these reasons, FAP is an attractive target and molecular imaging biomarker to assess CAFs and the tumour's landscape before and during immunotherapy. The PET radiotracer 68Ga-FAPI (Fibroblast activation protein inhibitor) allows the visualisation and quantification of CAFs.This study will use a non-invasive technique to assess CAFs before and during immunotherapy and to evaluate diverse predictive biomarkers in a prospective setting studying simultaneously CAFs (using 68Ga-FAPI) and cfDNA.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Pathologically- proven non-small-cell lung cancer (NSCLC).
* Proposed for treatment with anti-PD-(L)1 alone or in combination with chemotherapy and/or anti-CTLA4 in the advanced setting.
* ECOG Performance status ≤2.
* Patient's written informed consent obtained prior to any study procedure.

Exclusion Criteria:

* Surgery and/or radiotherapy to thoracic region within the last 8 weeks or anti-cancer systemic therapy within the last 2 weeks.
* Epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) and c-ros oncogene (ROS1) mutations.
* Pregnant and lactating women
* Previous or concurrent malignancy diagnosed within the last 2 years except adequately treated in situ carcinoma of the cervix uteri, localised (T1N0) low grade (Gleason score 6) prostate cancer undergoing active surveillance and basal or squamous cell skin cancer.
* Subjects with another significant medical condition which, in the investigator's opinion, may interfere with the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of inclusion until the date of first documented progression (RECIST) or date of death from any cause, whichever came first, assessed up to 24 months
  Patient outcome assessed by progression-free survival (PFS) defined as the time from the start of immunotherapy until disease progression* or death by any cause during the period of active and routine follow-up (overall PFS)

SECONDARY OUTCOMES:
Overall survival | until death by any cause, assessed up to 24 months
  Patient outcome assessed by 0verall survival (OS) defined as the time from the start of immunotherapy until death by any cause.
Objective response rate | From date of inclusion until the date of first documented progression (RECIST) or date of death from any cause, whichever came first, assessed up to 24 months
  Patient outcome assessed by objective response rate based on iRECIST criteria
  • Kinetics of imaging biomarkers assessed with 68Ga-FAPI PET/CT at baseline and during treatment - examples of kinetics of imaging biomarkers: ΔSUVmax / ΔSUVpeak / ΔUptake-Volume.
cfDNA | From date of inclusion until the date of last FAPI PET/CT (6 weeks after start immunotherapy)
  Kinetics of cfDNA values at baseline and during treatment
Number of lesions | From date of inclusion until the date of first documented progression (RECIST) or date of death from any cause, whichever came first, assessed up to 24 months
  Number of metastatic lesions and the imaging biomarkers (SUVmax / SUVpeak / Uptake-Volume / Tumour-to-Background ratio) of the lesions on 68Ga-FAPI PET/CT and 18F-FDG PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium